CLINICAL TRIAL: NCT06718699
Title: Accuracy of a New Prediction Equation to Calculate One Repetition Maximum (1RM) in Trained and Untrained Young and Old Adults
Brief Title: Accuracy of Prediction Equations to Calculate Maximum Strength
Status: Enrolling by invitation | Type: Observational
Sponsor: University of Erlangen-Nürnberg Medical School (Other)
Responsible Party: Principal Investigator, Wolfgang Kemmler, PhD, Professor Dr. PhD, Research Director, University of Erlangen-Nürnberg Medical School
Other Study IDs: PREDEQ; Physiomed ID 101 (Other: UKER - FAU)
Record Dates: First submitted 2024-12-01; First posted 2024-12-05 (Actual); Last update posted 2026-01-29 (Actual); Status verified 2026-01

CONDITIONS: Healthy Aging
Keywords: maximum strength; one repetition maximum; repetitions to fatigue; prediction equation; resistance exercise

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: resistance exercise tests — One 1RM and three RTF tests (5-8RM, 9-12RM, 13-16RM) on seven resistance training devices

SUMMARY:
Resistance exercise training (RT) is a key component of health related exercise programs. However, an accurate specification of RT load prescription is essential for effective and safe achievement of training aims. Proper specification of exercise intensity might be the most critical issue when designing RT protocols for adults. One repetition maximum tests (1RM) have been considered the "gold standard" of dynamic maximum strength evaluation. Although the argument of increased risk of injuries and adverse effects with 1RM testing in older people has been rejected by several studies , limited motivation to lift maximum loads, requirement for high test effort, time constraints, and interruption of the continuity of the training process aggravate the frequent application of 1RM tests particularly in non-athletic RT. 1RM prediction equations that use the load and number of repetitions completed to fatigue (RTF) to predict repetition maximum might be a reliable and feasible option to 1RM testing. Thus, the primary aims of this study were to evaluate the predictive accuracy of current RTF equations and to develop an equation that more accurately predicts 1RM from RTF tests.

ELIGIBILITY:
Inclusion Criteria:

* 18 to 35 years old
* 60 to 85 years old

Exclusion Criteria:

* Contraindication for one repetition maximum tests
* musculoskeletal injuries that may prevent a reliable and safe assessment of the 1RM and RTF tests

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The study population consists of resistance trained and untrained women and men 18 to 35 or 60-85 years old that are able to complete 1RM and RTF tests without endangering their health
Sampling Method: Non-Probability Sample
Enrollment: 120 (Estimated)
Dates: Start 2024-12-02 (Actual); Primary Completion 2026-08-31 (Estimated); Study Completion 2026-09-30 (Estimated)

PRIMARY OUTCOMES:
Maximum load, one repetition maximum, leg press | At baseline - no follow up tests
  Maximum load lifted once (1RM, in kg) for the leg press exercise

SECONDARY OUTCOMES:
Maximum load lifted at 5-8RM, leg press | At baseline - no follow up tests
  Maximum load lifted 5-8 times (RFT5-8, in kg) for the leg press exercise
Maximum load lifted at 9-12RM, leg press | At baseline - no follow up tests
  Maximum load lifted 5-8 times (RFT9-12, in kg) for the leg press exercise
Maximum load lifted at 13-16 RM, leg press | At baseline - no follow up tests
  Maximum load lifted 5-8 times (RFT13-16, in kg) for the leg press exercise
Maximum load, one repetition maximum, lat pulls | At baseline - no follow up tests
  Maximum load lifted once (1RM, in kg) for the latissimus pull exercise
Maximum load lifted at 5-8 RM, lat pulls | At baseline - no follow up tests
  Maximum load lifted 5-8 times (RFT5-8, in kg) for the latissimus pull exercise
Maximum load lifted at 9-12 RM, lat pulls | At baseline - no follow up tests
  Maximum load lifted 9-12 times (RFT9-12, in kg) for the latissimus pull exercise
Maximum load lifted at 13-16 RM, lat pulls | At baseline - no follow up tests
  Maximum load lifted 13-16 times (RFT13-16, in kg) for the latissimus pull exercise
Maximum load, one repetition maximum, triceps dips | At baseline - no follow up tests
  Maximum load lifted once (1RM, in kg) for the triceps dips exercise
Maximum load lifted at 5-8 RM, triceps dips | At baseline - no follow up tests
  Maximum load lifted 5-8 times (RFT5-8, in kg) for the triceps dips exercise
Maximum load lifted at 9-12 RM, triceps dips | At baseline - no follow up tests
  Maximum load lifted 9-12 times (RFT9-12, in kg) for the triceps dips exercise
Maximum load lifted at 13-16 RM, triceps dips | At baseline - no follow up tests
  Maximum load lifted 13-16 times (RFT13-16, in kg) for the triceps dips exercise
Maximum load, one repetition maximum, trunk extension | At baseline - no follow up tests
  Maximum load lifted once (1RM, in kg) for the trunk extension exercise
Maximum load lifted at 5-8 RM, trunk extension | At baseline - no follow up tests
  Maximum load lifted 5-8 times (RFT5-8, in kg) for the trunk extension exercise
Maximum load lifted at 9-12 RM, trunk extension | At baseline - no follow up tests
  Maximum load lifted 9-12 times (RFT9-12, in kg) for the trunk extension exercise
Maximum load lifted at 13-16 RM, trunk extension | At baseline - no follow up tests
  Maximum load lifted 13-16 times (RFT13-16, in kg) for the trunk extension exercise
Maximum load, one repetition maximum, trunk flexion | At baseline - no follow up tests
  Maximum load lifted once (1RM, in kg) for the trunk flexion exercise
Maximum load lifted at 5-8 RM, trunk flexion | At baseline - no follow up tests
  Maximum load lifted 5-8 times (RFT5-8, in kg) for the trunk flexion exercise
Maximum load lifted at 9-12 RM, trunk flexion | At baseline - no follow up tests
  Maximum load lifted 9-12 times (RFT9-12, in kg) for the trunk flexion exercise
Maximum load lifted at 13-16 RM, trunk flexion | At baseline - no follow up tests
  Maximum load lifted 13-16 times (RFT13-16, in kg) for the trunk flexion exercise
Maximum load, one repetition maximum, leg flexion | At baseline - no follow up tests
  Maximum load lifted once (1RM, in kg) for the leg flexion exercise
Maximum load lifted at 5-8 RM, leg flexion | At baseline - no follow up tests
  Maximum load lifted 5-8 times (RFT5-8, in kg) for the leg flexion exercise
Maximum load lifted at 9-12 RM, leg flexion | At baseline - no follow up tests
  Maximum load lifted 9-12 times (RFT9-12, in kg) for the leg flexion exercise
Maximum load lifted at 13-16 RM, leg flexion | At baseline - no follow up tests
  Maximum load lifted 13-16 times (RFT13-16, in kg) for the leg flexion exercise
Maximum load, one repetition maximum, leg extension | At baseline - no follow up tests
  Maximum load lifted once (1RM, in kg) for the leg extension exercise
Maximum load lifted at 5-8 RM, leg extension | At baseline - no follow up tests
  Maximum load lifted 5-8 times (RFT5-8, in kg) for the leg extension exercise
Maximum load lifted at 9-12 RM, leg extension | At baseline - no follow up tests
  Maximum load lifted 9-12 times (RFT9-12, in kg) for the leg extension exercise
Maximum load lifted at 13-16 RM, leg extension | At baseline - no follow up tests
  Maximum load lifted 13-16 times (RFT13-16, in kg) for the leg extension exercise

CONTACTS AND LOCATIONS:
Locations (1):
- Institute of Radiology, University Hospital NErlangen, Erlangen, Germany